CLINICAL TRIAL: NCT01815840
Title: A Randomized, Double-blinded, Regimen-controlled, Phase II, Multicenter Study to Assess the Efficacy and Safety of Two Different Vismodegib Regimens in Patients With Multiple Basal Cell Carcinomas
Brief Title: A Study of Two Vismodegib Regimens in Participants With Multiple Basal Cell Carcinomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MO28295; 2012-003305-10 (EudraCT Number)
Record Dates: First submitted 2013-03-19; First posted 2013-03-21 (Estimated); Results first posted 2016-08-04 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-08

CONDITIONS: Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — HhAntag691

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vismodegib Intermittent Schedule (Experimental): Vismodegib intermittent schedule of 12 weeks vismodegib followed by 8 weeks placebo, repeated 3 times with a final course of vismodegib (total 72 weeks), followed by 52 weeks treatment-free follow up
  Interventions: Drug: Vismodegib; Drug: Placebo
- Vismodegib Induction Followed by Intermittent Schedule (Experimental): Vismodegib beginning with 24 weeks induction followed by intermittent schedule 8 weeks placebo, 8 weeks vismodegib (total 72 weeks), followed by 52 weeks treatment-free follow up
  Interventions: Drug: Vismodegib; Drug: Placebo

INTERVENTIONS:
Drug: Vismodegib — Vismodegib 150 mg hard gelatin capsule orally once daily
  Other Names: Erivedge®
Drug: Placebo — Vismodegib placebo orally once daily

SUMMARY:
This randomized, double-blind, regimen-controlled, phase II, multicenter study will assess the efficacy and safety of two different vismodegib regimens in participants with multiple basal cell carcinoma. Participants will receive vismodegib 150 mg orally once daily either in an intermittent schedule of 12 weeks vismodegib followed by 8 weeks placebo (Arm A) or as 24 weeks induction followed by an intermittent schedule of 8 weeks placebo followed by 8 weeks vismodegib (Arm B). Anticipated time on study treatment is 72 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, >/= 18 years of age
* Participants with multiple basal cell carcinomas, including participants with Gorlin syndrome, with at least 6 clinically evident basal cell carcinomas at the time of randomization, of which 3 measure 5 mm or more in diameter and are considered target lesions. All other lesions are considered to be non-target lesions
* Histopathologic confirmation that at least one of the three target lesions is basal cell carcinoma
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Adequate renal and hepatic function and hematopoietic capacity
* Women of childbearing potential must agree to use contraception as defined by protocol during treatment and for at least 9 months after completion of study treatment
* Male participants with female partners of childbearing potential must agree to use contraception as defined by protocol during treatment and for 2 months after completion of study treatment

Exclusion Criteria:

* Inability or unwillingness to swallow capsules
* Pregnant or breastfeeding women
* Any metastatic basal cell carcinoma
* Locally advanced basal cell carcinoma lesion that is considered to be inoperable or to have medical contraindications to surgery
* Recent (i.e., within the past 28 days prior to randomization) or current participation in another experimental drug study
* Known or suspected alcohol abuse
* One of the following known rare hereditary conditions: galactose intolerance, primary hypolactasia or glucose-galactose malabsorption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2013-04-30 (Actual); Primary Completion 2015-08-27 (Actual); Study Completion 2016-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (58):
- United States (17):
  - Dermatology Research Associate, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Skin Surgery Med Group, Inc, San Diego, California
  - California Pacific Medical Center Research Institute, Santa Rosa, California
  - Advanced Derm & Cosmetic Surg, Ormond Beach, Florida
  - Skin and Cancer Associates and the Center for Cosmetic Enhancement, Plantation, Florida
  - Emory University Clinic, Atlanta, Georgia
  - Laser & Skin Surgery Center of Indiana, Carmel, Indiana
  - Beverly Hospital;Oncology Center Pharmacy, Beverly, Massachusetts
  - Saint Louis University School of Medicine; Department of Dermatology, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Long Island Skin Cancer and Dermatologic Surgery, Smithtown, New York
  - Mariwalla Dermatology, West Islip, New York
  - The Skin Surgery Center, Winston-Salem, North Carolina
  - Ohio State University, Columbus, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Dermatology and Laser Center of Charleston PA, Charleston, South Carolina
- Austria (2):
  - LKH Innsbruck; Universitätsklinik für Dermatologie, Innsbruck
  - Medizinische Universität Wien; Univ.Klinik für Dermatologie, Vienna
- Canada (3):
  - UBC Department of Dermatology & Skin Sciences, Vancouver, British Columbia
  - Dermetics, Burlington, Ontario
  - Innovaderm Research Inc., Montreal, Quebec
- France (10):
  - CHU Amiens - Hopital Sud, Amiens
  - Hopital Saint Andre CHU De Bordeaux; Dermatologie, Bordeaux
  - Chu Site Du Bocage;Dermatologie, Dijon
  - Hopital Dupuytren; Dermatologie, Limoges
  - Hopital Timone Adultes; Dermatologie, Marseille
  - Hopital Saint Eloi; CHU de Montpellier; Svc de Dermatologie, Montpellier
  - Hopital Hotel Dieu Et Hme; Clinique Dermatologique, Nantes
  - Hôpital Saint-Louis, Paris
  - Ch Francois Mitterrand; Medecine Oncologie, Pau
  - Hopital Nord ; Dermatologie, Saint-Etienne
- Germany (8):
  - Universitätsklinik Essen; Klinik und Poliklinik für Dermatologie, Venerologie und Allergologie, Essen
  - Klinik Johann Wolfgang von Goethe Uni; Klinik für Dermatologie, Venerologie und Allergologie, Frankfurt
  - SRH Wald-Klinikum Gera; Klinik für Hautkrankheiten und Allergologie, Gera
  - Medizinische Hochschule Hannover; Klinik für Dermatologie, Allergologie und Venerologie, Hanover
  - UNI-Klinikum Campus Kiel Klinik f.Dermatologie Tagesklinik f.Dermatologie, Kiel
  - Klinikum der LMU München; Klinik und Poliklinik für Dermatologie und Allergologie, München
  - Fachklinik Hornheide; Dermatologie, Münster
  - Universitätsklinikum Tübingen Universitäts-Hautklinik, Tübingen
- Italy (5):
  - Ospedale San Salvatore (ASL-01); Dip. di Dermatologia U.O.S. di Dermatologia Oncol, L’Aquila, Abruzzo
  - Arcispedale Santa Maria Nuova; Dermatologia, Reggio Emilia, Emilia-Romagna
  - Università di Brescia; Dipartimento di Dermatologia, Brescia, Lombardy
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Turin, Piedmont
  - Ospedale IOT- Palagi Dermatologia 2, Florence, Tuscany
- Mexico (2):
  - Hospital General de México, Mexico City
  - Hospital General Dr. Manuel Gea Gonzalez; Dermatology, México
- Netherlands (3):
  - VU MEDISCH CENTRUM;Afdeling Dermatologie, Amsterdam
  - Academ Ziekenhuis Groningen; Medical Oncology, Groningen
  - Maastricht University Medical Centre; Dermatologie, Maastricht
- Russia (3):
  - Blokhin Cancer Research Center; General Oncology Department, Moscow
  - FSBI "Russian Oncology Research Center n.a. N. N. Blokhin" of Ministry of Health of the Russian Fed, Moscow
  - City Clinical Oncology Dispensary, Saint Petersburg
- Spain (5):
  - Hospital Costa Del Sol; Servicio de Dermatologia, Málaga, Malaga
  - Hospital Clinic i Provincial; Servicio de Farmacia, Barcelona
  - Hospital General Universitario de Guadalajara; Servicio de Dermatologia, Guadalajara
  - Hospital General Universitario de Valencia; Servicio de oncologia, Valencia
  - Instituto Valenciano Oncologia; Oncologia Medica, Valencia

REFERENCES:
- [Derived] Jacobsen AA, Kydd AR, Strasswimmer J. Practical management of the adverse effects of Hedgehog pathway inhibitor therapy for basal cell carcinoma. J Am Acad Dermatol. 2017 Apr;76(4):767-768. doi: 10.1016/j.jaad.2016.04.063. No abstract available. PMID 28325399
- [Derived] Dreno B, Kunstfeld R, Hauschild A, Fosko S, Zloty D, Labeille B, Grob JJ, Puig S, Gilberg F, Bergstrom D, Page DR, Rogers G, Schadendorf D. Two intermittent vismodegib dosing regimens in patients with multiple basal-cell carcinomas (MIKIE): a randomised, regimen-controlled, double-blind, phase 2 trial. Lancet Oncol. 2017 Mar;18(3):404-412. doi: 10.1016/S1470-2045(17)30072-4. Epub 2017 Feb 8. PMID 28188086

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 229 participants were enrolled in 10 countries.
Period: Overall Study
Arm/Group | Vismodegib Intermittent Schedule | Vismodegib Induction Followed by Intermittent Schedule
Started | 116 | 113
Completed | 57 | 50
Not Completed | 59 | 63
Not completed — Missing | 1 | 0
Not completed — Withdrew Consent | 31 | 30
Not completed — Administrative/Other | 1 | 3
Not completed — Adverse Event | 10 | 16
Not completed — Death | 2 | 2
Not completed — Disease progression | 3 | 2
Not completed — Investigators Decision | 2 | 3
Not completed — Lost to Follow-up | 3 | 6
Not completed — Refused Treatment | 5 | 1
Not completed — Sponsor Termination Treatment | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Analysis Population, defined as all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vismodegib Intermittent Schedule | Vismodegib Induction Followed by Intermittent Schedule | Total
Number analyzed (Participants) | 116 | 113 | 229
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (13.94) | 59.9 (15.35) | 60.5 (14.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 25 | 60
  Male | 81 | 88 | 169

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change From Baseline in the Number of Clinically Evident Basal Cell Carcinomas at Week 73 (After 72 Weeks of Treatment)
Description: The total number of clinically evident basal cell carcinomas = the total number of target and/or non-target lesions present in individual participants.
Time Frame: Baseline; Week 73
Population: Participants in the Intent-to-Treat analysis population (defined as all randomized participants) with available data were included in the analysis. The last observation carried forward method was used.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Vismodegib Intermittent Schedule | Vismodegib Induction Followed by Intermittent Schedule
Number analyzed (Participants) | 114 | 113
percent change | 62.9 (52.01) | 54.9 (54.85)
Statistical Analysis 1: Comparison: Vismodegib Intermittent Schedule vs Vismodegib Induction Followed by Intermittent Schedule; The mean difference in the mean relative reduction between treatment arms, along with the corresponding 95% confidence interval, was estimated by fitting an ANCOVA model with treatment as main effect and the following covariates: number of basal cell carcinomas at baseline, geographical region, immunosuppression status, confirmed basal cell carcinoma nevus syndrome; Test type: Superiority or Other; Mean Difference (Final Values) = -8.3, 95% CI 2-sided [-22.2 to 5.7] — Asymptotic confidence intervals are presented for the difference between treatment arms

2. Secondary Outcome: Percentage of Participants Who Discontinued Study Treatment Due to Tolerability Issues
Description: The percentage of participants who discontinued study treatment (due either to adverse event, refusal of treatment, or withdrawal of consent) was summarized by treatment group.
Time Frame: Baseline to Week 73
Population: Intent-to-Treat Analysis Population, defined as all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vismodegib Intermittent Schedule | Vismodegib Induction Followed by Intermittent Schedule
Number analyzed (Participants) | 116 | 113
percentage of participants
  Overall | 37.1 [28.3 to 46.5] | 41.6 [32.4 to 51.2]
  Adverse Events | 20.7 [13.7 to 29.2] | 27.4 [19.5 to 36.6]
  Refused Treatment | 6.0 [2.5 to 12.0] | 2.7 [0.6 to 7.6]
  Withdrew Consent | 10.3 [5.5 to 17.4] | 11.5 [6.3 to 18.9]

3. Secondary Outcome: Mean Percent Change From Baseline in Total Size of Three Target Basal Cell Carcinoma Lesions in Individual Participants at Week 73
Description: The three target basal cell carcinoma lesions = the three largest visible lesions, at least 5 mm in the longest diameter, in individual participants.
Time Frame: Baseline; Week 73
Population: Participants in the Intent-to-Treat Analysis Population (defined as all randomized participants) with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Vismodegib Intermittent Schedule | Vismodegib Induction Followed by Intermittent Schedule
Number analyzed (Participants) | 94 | 86
percent change | 82.9 (27.01) | 68.0 (53.02)

4. Secondary Outcome: Percentage of Participants With at Least 50% Reduction in the Number of Basal Cell Carcinomas at Week 73
Time Frame: Baseline; Week 73
Population: Intent-to-Treat Analysis Population, defined as all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Vismodegib Intermittent Schedule | Vismodegib Induction Followed by Intermittent Schedule
Number analyzed (Participants) | 116 | 113
percentage of participants | 65.5 | 50.4

5. Secondary Outcome: Percentage of Participants With New Basal Cell Carcinomas at Week 73
Time Frame: Baseline; Week 73
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Vismodegib Intermittent Schedule | Vismodegib Induction Followed by Intermittent Schedule
Number analyzed (Participants) | 94 | 86
percentage of participants
  No new lesions | 76.6 | 74.4
  1 new lesion | 10.6 | 11.6
  2 new lesions | 5.3 | 5.8
  3 new lesions | 5.3 | 2.3
  >3 new lesions | 2.1 | 5.8

6. Secondary Outcome: Percent Change in Total Number of Basal Cell Carcinomas Relative to Baseline at Week 85 (12 Weeks Following End of Treatment) (Recurrence Rate)
Time Frame: Baseline; Week 85
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Vismodegib Intermittent Schedule | Vismodegib Induction Followed by Intermittent Schedule
Number analyzed (Participants) | 90 | 77
percent change | 35.7 (50.25) | 38.5 (55.22)

7. Secondary Outcome: Percent Change in Total Number of Basal Cell Carcinomas Relative to Baseline at Week 97 (24 Weeks Following End of Treatment) (Recurrence Rate)
Time Frame: Baseline; Week 97
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Vismodegib Intermittent Schedule | Vismodegib Induction Followed by Intermittent Schedule
Number analyzed (Participants) | 84 | 72
percent change | 36.0 (49.48) | 42.1 (57.83)

8. Secondary Outcome: Percent Change in Total Number of Basal Cell Carcinomas Relative to Baseline at Week 125 (52 Weeks Following End of Treatment) (Recurrence Rate)
Time Frame: Baseline; Week 125
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Vismodegib Intermittent Schedule | Vismodegib Induction Followed by Intermittent Schedule
Number analyzed (Participants) | 95 | 82
percent change | 41.2 (45.23) | 44.0 (42.87)

9. Secondary Outcome: Percentage of Participants Experiencing Any Adverse Event
Time Frame: Up to 125 weeks
Population: Safety Analysis Population: participants in the Intent-to-Treat Analysis Population (defined as all randomized participants) who received at least one dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Vismodegib Intermittent Schedule | Vismodegib Induction Followed by Intermittent Schedule
Number analyzed (Participants) | 114 | 113
percentage of participants | 99.1 | 97.3

10. Secondary Outcome: Percent Change From Baseline in the Skindex-16 Symptom Domain Score at Week 73
Description: The Skindex-16 is a patient-reported outcome health questionnaire. Participants were asked about their symptoms, and their answers were combined into a composite Symptom Domain Score. Scores range from 0 ("never bothered") to 100 ("always bothered").
Time Frame: Baseline; Week 73
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Vismodegib Intermittent Schedule | Vismodegib Induction Followed by Intermittent Schedule
Number analyzed (Participants) | 87 | 79
percent change | -14.9 (25.75) | -12.6 (23.98)

11. Secondary Outcome: Percent Change From Baseline in the Skindex-16 Emotion Domain Score at Week 73
Description: The Skindex-16 is a patient-reported outcome health questionnaire. Participants were asked about their emotional state, and their answers were combined into a composite Emotion Domain Score. Scores range from 0 ("never bothered") to 100 ("always bothered").
Time Frame: Baseline; Week 73
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Vismodegib Intermittent Schedule | Vismodegib Induction Followed by Intermittent Schedule
Number analyzed (Participants) | 87 | 79
percent change | -27.4 (27.71) | -28.9 (28.16)

12. Secondary Outcome: Percent Change From Baseline in the Skindex-16 Function Domain Score at Week 73
Description: The Skindex-16 is a patient-reported outcome health questionnaire. Participants were asked about their ability to function, and answers were combined into a composite Function Domain Score. Scores range from 0 ("never bothered") to 100 ("always bothered").
Time Frame: Baseline; Week 73
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Vismodegib Intermittent Schedule | Vismodegib Induction Followed by Intermittent Schedule
Number analyzed (Participants) | 87 | 79
percent change | -9.5 (20.59) | -10.3 (26.03)

ADVERSE EVENTS:
Time Frame: Up to 125 weeks
Description: Safety Analysis Population: participants in the Intent-to-Treat Analysis Population (defined as all randomized participants) who received at least one dose of study treatment.
Arm/Group | Vismodegib Intermittent Schedule | Vismodegib Induction Followed by Intermittent Schedule
Serious Adverse Events (participants affected / at risk) | 24/114 | 23/113
Other Adverse Events (participants affected / at risk) | 107/114 | 108/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vismodegib Intermittent Schedule (N=114) | Vismodegib Induction Followed by Intermittent Schedule (N=113)
Pneumonia (Infections and infestations) | 3 | 0
Abscess limb (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 1
Kidney infection (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Spindle cell sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1
Nervous system disorder (Nervous system disorders) | 0 | 1
Post herpetic neuralgia (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pseudolymphoma (Blood and lymphatic system disorders) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
International normalized ratio increased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Personality change (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1
Congenital cerebral cyst (Congenital, familial and genetic disorders) | 1 | 0
Asthenia (General disorders) | 1 | 1
Acute hepatic failure (Hepatobiliary disorders) | 0 | 1
Primary amyloidosis (Immune system disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Xanthelasma (Skin and subcutaneous tissue disorders) | 1 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Haematoma (Vascular disorders) | 0 | 1
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vismodegib Intermittent Schedule (N=114) | Vismodegib Induction Followed by Intermittent Schedule (N=113)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 83 | 94
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 16
Myalgia (Musculoskeletal and connective tissue disorders) | 18 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 7
Dysgeusia (Nervous system disorders) | 76 | 75
Ageusia (Nervous system disorders) | 13 | 14
Headache (Nervous system disorders) | 10 | 14
Alopecia (Skin and subcutaneous tissue disorders) | 72 | 73
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 13
Actinic keratosis (Skin and subcutaneous tissue disorders) | 10 | 8
Diarrhoea (Gastrointestinal disorders) | 20 | 20
Nausea (Gastrointestinal disorders) | 23 | 14
Abdominal pain (Gastrointestinal disorders) | 8 | 12
Constipation (Gastrointestinal disorders) | 9 | 8
Abdominal pain upper (Gastrointestinal disorders) | 9 | 5
Vomiting (Gastrointestinal disorders) | 7 | 4
Fatigue (General disorders) | 24 | 26
Asthenia (General disorders) | 15 | 21
Weight decreased (Investigations) | 24 | 21
Blood creatine phosphokinase increased (Investigations) | 11 | 15
Alanine aminotransferase increased (Investigations) | 7 | 5
Nasopharyngitis (Infections and infestations) | 7 | 12
Folliculitis (Infections and infestations) | 10 | 8
Bronchitis (Infections and infestations) | 5 | 8
Upper respiratory tract infection (Infections and infestations) | 7 | 5
Decreased appetite (Metabolism and nutrition disorders) | 21 | 17
Eczema (Skin and subcutaneous tissue disorders) | 6 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 7
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 6 | 2
Insomnia (Psychiatric disorders) | 5 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Hypertension (Vascular disorders) | 2 | 6
Pyrexia (General disorders) | 1 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.